CLINICAL TRIAL: NCT01931488
Title: The Feasibility of Novel 124I-MIBG Tracer in Evaluation of Myocardial Sympathetic Denervation and Assessment of Neuroendocrine Tumors. Comparison With 123I-MIBG.
Brief Title: 124I-MIBG Tracer Evaluation of Myocardial Sympathetic Denervation and Assessment of Neuroendocrine Tumors.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, DIRECTOR, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-12-ES-0341-CTIL
Record Dates: First submitted 2013-08-14; First posted 2013-08-29 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Parkinson Disease; Neuroendocrine Tumors
MeSH Terms: conditions — Parkinson Disease; Neuroendocrine Tumors | interventions — Iodine-123; Iodine-124; Tomography, Emission-Computed, Single-Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MIBG label with I123 or I124 (Other): evaluate the added value of PET-CT with 124I-MIBG tracer, compared to planar and SPECT imaging with the routine 123I-MIBG tracers/
  Interventions: Other: MIBG label with I123 or I124; Device: SPECT imaging

INTERVENTIONS:
Other: MIBG label with I123 or I124 — PD Patients who are not allergic to Iodine will be given 8 drops of Lugol . 30 min later, patients will be injected with 123I-MIBG 6 mci (222 MBq). 3 hours post-injection patients will undergo planar and SPECT imaging. at another day, patients will be injected with 124I-MIBG 0.8 mci (29.6 MBq). 3 hours post-injection patients will undergo PET-CT imaging.whole-body imaging. in the evaluation of neuroendocrine tumors-Patients who are not allergic to Iodine will be given 8 drops of Lugol.30 min later, patients will be injected with 123I-MIBG 6 mCi (222 MBq).3 hours and 24 hours post-injection patients will undergo planar and SPECT imaging. at another day, patients will be injected with 124I-MIBG 0.8 mCi (29.6 MBq). 3 hours and 24 hours post-injection patients will undergo PET-CT imaging.
Device: SPECT imaging

SUMMARY:
The Feasibility of Novel 124I-MIBG Tracer in Evaluation of Myocardial Sympathetic Denervation and Assessment of Neuroendocrine tumors. Comparison with 123I-MIBG.

DETAILED DESCRIPTION:
The autonomic nervous system consists of sympathetic and parasympathetic innervation.

The neurotransmitter of the sympathetic system is norepinephrine (NE) which in response to a stimulus, is released to the synaptic space Guanethidine is a false neurotransmitter analog of NE that is not catabolized . When labeled with radioactive iodine the radiotracer meta-iodobenzylguanidine (as I-MIBG) may be used for localization of different clinical and pathological conditions. There are two main indications for scintigrpahy with labeled MIBG 1. Whole body imaging of neuroendocrine tumors such as phechromocytoma and neuroblastoma. Scintigraphy allows staging of the disease as well as follow up in patients with MIBG-avid tumors. Moreover, when labeled with high doses of 131I it can be used for treatment in patients with metastatic neuroendocrine tumors. 2. the other indication of labeled MIBG scintigraphy is for assessment of myocardial sympathetic nerve endings Autonomic disturbances are of the common symptoms in Parkinson disease (PD). They may appear early in the disease occasionally prior to the motor symptoms, thus raising a potential use of autonomic system assessment as a biological marker for prediction of future development of motor PD.

Labeled MIBG imaging is a potential test for determining of the integrity of the individual autonomic function. Reduced MIBG uptake indicates postganglionic sympathetic dysfunction, which has been observed during the early stages of PD. MIBG scintigraphy is thought to be a sensitive modality for the diagnosis of PD, assisting in the differential diagnosis of other parkinsonian diseases, PD and other movement disorders. This method has also been reported to be of a high specificity.

The labeled MIBG used routinely is the tracer labeled with 123I which can be used with gamma camera for performance of planar imaging or 3D SPECT images. 123I emits predominantly γ photons with energies of 159 keV and has a half-life of 13.2 hour.

Quantitation of 123I MIBG myocardial uptake by the Heart to-Mediastinum ratio (H/M) measured from planar imaging has been found to be of predictive value for assessment of prognosis for cardiac events. H/M obtained from 123I MIBG SPECT was reported to improve the differentiation between subjects with normal and those with abnormal MIBG uptake.

Unlike 123I which is a gamma emitting isotope 124I, a positron emitter, with a half-life of 4.2 d, can be used for positron emission tomography (PET) thus allowing a better as well as quantification of tracer accumulation Studies using 124I-MIBG positron emission tomography was initiated as early as 1992. Preliminary studies demonstrated that imaging with 124I-MIBG in humans is safe when using the correct amount of radioactivity tracer.

In this study we propose to perform two images sessions. First would be the injection of 6mCi 123I-MIBG which results in radiation dose of 4.2 mSv.In the second session 0.8 mCi 124I-MIBG will be injected which results in radiation dose of 7.4 mSv. The estimated total radiation dose to the patient of both studies is 11.8 mSv. When comparing to the radiation doses of daily routine scintigraphy: The radiation dose of bone scan (25 mCi Tc MDP) is 5.3 mSv. The radiation dose of 12 mCi 18F-FDG PET-CT is 13.32 mSv.

Trail Objectives Given the merits of MIBG ligand and the 124I positron emission tomography, the purpose of this study is to evaluate the added value of PET-CT with 124I-MIBG tracer, compared to planar and SPECT imaging with the routine 123I-MIBG tracers for

1. Assessment of the Myocardial Sympathetic Denervation of patients with Parkinson and family members of patienst with PD who are carriers of the mulation for PD.
2. Staging and follow-up of pts. with neuroendocrine malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Signed Informed Consent
* Patients diagnosed with Parkinson disease
* Patients with histologically confirmed neuroendocrine tumors

Exclusion Criteria:

* Age < 18
* Any cardiovascular disease
* Taking medications that influence the sympathetic system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Uptake of 123I-MIBG | day 1
  At day 1 patients will be injected with 123I-MIBG 6 mci (222 MBq). 3 hours post-injection patients will undergo planar and SPECT imaging. Uptake of 123I-MIBG will be quantified as heart/mediastinum ratio measured from planar imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Einat Even Sapir, PhD, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel, Israel